CLINICAL TRIAL: NCT05106452
Title: Intraoperative Analgesia Management in Gynecological Surgery With Erector Spinae Block
Brief Title: Effect of ANI on Intraoperative Opioid Consumption
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zonguldak Bulent Ecevit University (Other)
Collaborators: Zeynep Koc (Unknown)
Responsible Party: Principal Investigator, Çağdaş Baytar, assistant professor, Zonguldak Bulent Ecevit University
Other Study IDs: 2021/18-4
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Analgesia; Nociceptive Pain; Nerve Block; Pain
Keywords: Analgesia nociception index; Pain monitoring; Analgesia
MeSH Terms: conditions — Agnosia; Nociceptive Pain; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group ANI
- Group Control

SUMMARY:
The aim of the study is to compare the analgesic nociception index (ANI), which is used to determine the dose of analgesic agent needed in the intraoperative period, with the conventional method in patients with erector spinae block who underwent gynecological surgery under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II-III risk group
* Patients who underwent gynecological surgery under general anesthesia, who underwent erector spina block, and whose pain was followed by analgesia nociception index or conventional methods for intraoperative pain monitoring
* Patients whose informed consent was read and consent was obtained from them and their guardians

Exclusion Criteria:

* cardiac rhythm disorder
* central-autonomic nervous system disease
* neuropsychiatric disease
* receiving opioid therapy
* Use of drugs that will affect cardiac autonomic regulation
* Known allergy to the drugs to be applied
* Contraindicated for ESP block
* Patients who do not agree to participate in the study will not be included in the study.
* Patients who were administered drugs to stabilize the patient's hemodynamics during the operation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: female patients gynecological surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
intraoperative opioid consumption | during the surgery
  Effect of ANI monitoring on intraoperative opioid consumption

SECONDARY OUTCOMES:
emergence time | at the end of the surgery
  time between last suture and extubation
VAS pain scores | during her stay in the recovery unit
  pain scores in the recovery unit
duration of stay in recovery room | at the end of the surgery
  time between entering and exiting the recovery unit
nausea and vomiting i | during her stay in the recovery unit
  incidence of nausea and vomiting in recovery room

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University Medicine Faculty, Zonguldak, Kozlu, Turkey (Türkiye)

REFERENCES:
- [Derived] Koc Z, Baytar C, Bollucuoglu K, Koksal BG, Okyay RD, Piskin O, Ayoglu H. Intraoperative analgesia management by monitoring the analgesia nociception index in gynecological surgeries involving erector spinae plane block: a randomized controlled study. J Clin Monit Comput. 2025 Dec;39(6):1185-1191. doi: 10.1007/s10877-025-01330-x. Epub 2025 Jul 15. PMID 40663304